CLINICAL TRIAL: NCT04029259
Title: Evaluation of Pre- and Post-operative Brain MRI in Carotid Endarterectomy
Brief Title: Pre- and Post-operative Brain MRI in Carotid Endarterectomy
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Toril Rabben, Consultant in Vascular Surgery, Oslo University Hospital
Other Study IDs: MR caput and CEA
Record Dates: First submitted 2017-08-03; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Carotid Artery Stenoses
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Brain MRI — Brain MRI diagnoses tromboembolic lesions or bleeding to the cerebrum and is part of preoperative diagnostic tests before carotid surgery. After surgery brain MRI may present New lesions related to surgery, clinically significant or insignificant. Our goal is to evaluate the relevance of this modality in carotid surgery..

SUMMARY:
Patients undergoing carotid endarterectomy in the Department of Vascular Surgery at Oslo University Hospital are consecutively included in this evaluation og pre- and postoperative brain MRI.

DETAILED DESCRIPTION:
Patients undergoing surgery for carotid stenosis in our Department are examined by brain MRI before and after carotid surgery to evaluate the rationale for the MRI. Brain lesions on MRI before and after carotid surgery are registered, and related to clinical findings. The purpose of the study is to evaluate whether brain MRI in relation to carotid endarterectomy gives additional information to clinical findings, and to CT scan of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Indication for carotid surgery

Exclusion Criteria:

* Contraindications to MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to the Department of Vascular Surgery at Oslo University Hospital for carotid endarterectomy. International guidelines on indications for surgery are followed, and the majority of the patients have symptomatic carotid stenosis occluding > 70% of the lumen of the internal carotid artery. Patients characteristics and indications for surgery are registered
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Brain lesions on MRI | 30 days
  Lesions on brain MRI representing thromboembolic or hemorrhagic episodes

SECONDARY OUTCOMES:
Time from Transient Ischemic Attack (TIA) or minor stroke to surgery | Days before surgery, maximum 6 months
  International guidelines recommends surgery within 14 days after TIA

OTHER OUTCOMES:
Complications to carotid surgery | Within 30 days after surgery
  TIA, minor stroke, nerve damage

CONTACTS AND LOCATIONS:
Overall Officials: Toril Rabben, PhD, Principal Investigator — Oslo University Hospital, Dep. of Vascular Surgery

IPD SHARING:
Plan to Share IPD: Undecided
No plan